CLINICAL TRIAL: NCT03700359
Title: A Randomized, Open-label Study of Lobaplatin/Etoposide as First Line Therapy With or Without Anlotinib Maintenance Therapy in Patients With Extensive-stage Small-cell Lung Cancer
Brief Title: A Study of Lobaplatin/Etoposide With or Without Anlotinib Maintenance Therapy in Patients With ES-SCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jiexia Zhang, Deputy Director, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ES-SCLC 001
Record Dates: First submitted 2018-07-29; First posted 2018-10-09 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Small Cell Lung Carcinoma
Keywords: extensive-stage small-cell lung cancer; lobaplatin/etoposide; Anlotinib maintenance therapy
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — anlotinib; lobaplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anlotinib/Lobaplatin/Etoposide (Experimental): EL regimen for 4 cycles followed by Anlotinib Hydrochloride maintenance therapy
  Interventions: Drug: Anlotinib Hydrochloride; Drug: Lobaplatin; Drug: Etoposide
- Lobaplatin/Etoposide (Active Comparator): EL regimen for 4 cycles
  Interventions: Drug: Lobaplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Anlotinib Hydrochloride — Anlotinib: Maintenance therapy 12mg/day P.O., day 1-15 every 21 days (2 weeks on, 1 week off) until progressive disease or treatment discontinuation
  Other Names: AL3818
  Arms: Anlotinib/Lobaplatin/Etoposide
Drug: Lobaplatin — Lobaplatin:30 mg/m2 IV every 21 days for up to 4 cycles of 21 days
  Other Names: D-19466
Drug: Etoposide — Etoposide: 60 mg/m2 IV every 21 days for up to 4 cycles of 21 days
  Other Names: VP16

SUMMARY:
This is a prospective, randomized, open-label and active controlled phase II study. It plans to enroll 60 subjects with extensive stage small cell lung cancer (ES-SCLC). All subjects will be assigned randomly to the experimental arm or control arm. The primary endpoints would be overall survival and progression-free survival.

DETAILED DESCRIPTION:
Small cell lung cancer (SCLC) accounts for about 20% of lung cancer, has a high degree of malignancy, short doubling time, early and widespread metastasis, is sensitive to chemotherapy and radiotherapy, and has a high initial response rate, but is prone to secondary drug resistance and relapse. The treatment is mainly based on systemic chemotherapy.

SCLC has a more abundant vascular network than NSCLC. Anti-tumor vascular therapy combined with chemotherapy is considered the most promising SCLC first-line anti-tumor strategy. Anlotinib Hydrochloride has an anti-angiogenic effect and inhibits tumor's growth. It has been reported that Anlotinib has the dual benefits of both overall survival and progression-free survival in the treatment of multiple tumors, and has initially demonstrated its safety and efficacy. The ALTER 0303 study results showed that Anlotinib benefited both the overall and progression-free survival of NSCLC patients. However, there is no clinical study to probe its relevance to small cell lung cancer, and few studies have examined the status of Anlotinib in first-line treatment.

This randomized, open-label, controlled study is to evaluate the efficacy and safety of sequential EL regimen with Anlotinib hydrochloride as first-line treatment for extensive-stage SCLC. The study plan to enroll 60 ES-SCLC subjects and will provide evidence for the use of Anlotinib for SCLC first-line treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed patients with extensive small cell lung cancer;
2. Karnofsky performance status ≥70;
3. At least one lesion that can measured by CT;
4. Expected to survive for at least 3 months;
5. Peripheral blood and liver and kidney function within the following allowable range (tested within 7 days before treatment);

   * White blood cell (WBC) ≥3.0×109/L or Neutrophils (ANC) ≥1.5×109/L;
   * Hemoglobin (HGB) ≥80 g/L；
   * Platelet (PLT) ≥100×109/L;
   * Liver transaminases（AST/ALT）<3.0 times the normal range limit;
   * Total bilirubin（TBIL）<1.5 times the normal range limit;
   * Creatinine（CREAT）<1.5 times the normal range limit;
6. Patients of childbearing age (including female and male patients' partner) must take effective contraception methods;
7. Signed informed consent;
8. Known history of liver disease: Hepatitis B Virus (HBV) infection and Hepatitis B Virus DNA (HBV DNA ≥500 copies or ≥100 IU/ml); or Hepatitis C Virus (HCV) infection; or liver cirrhosis, etc.
9. Human immunodeficiency virus (HIV);
10. Subjects with difficulties in swallowing or known drug malabsorption; Those who meet each of the above criteria are included in the study.

Exclusion Criteria:

1. Other pathological types of tumor except for small cell lung cancer;
2. Patients with a history of severe allergies or allergies;
3. Pregnancy or breastfeeding women;
4. Patients who have previously participated in other clinical trials and have not yet terminated the trial;
5. Combined with other tumors at the time of initial diagnosis;
6. Patients who have previously participated in other clinical trials and have not yet terminated the trial;
7. Patients who have acute infection that difficult to control;
8. Drug abuse, substance abuse, chronic alcohol abuse, and AIDS patients. Those who meet any of the above criteria are not included in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-11-29 (Estimated); Study Completion 2021-11-29 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival Time | Time from randomization to first documented progression, assessed for up to 2 years
  Progression free survival (PFS) is defined as the time from date of randomization to the date of objective disease progression or death due to any cause. Participants were censored at date of last PFS assessment prior to the cutoff date or the date of initiation of subsequent systemic anticancer therapy, whichever was earlier.

SECONDARY OUTCOMES:
Percentage of Participants With a Complete Response (CR) and Partial Response (PR) (Overall Response Rate) | Up to 2 years
  Overall Response Rate (ORR) is the number of participants with a Complete Response (CR) and Partial Response (PR) divided by the total number of randomized participants per arm, then multiplied by 100. Response is based on the Response Evaluation Criteria In Solid Tumors (RECIST 1.0) criteria. Complete Response (CR) was defined as the disappearance of all target lesions. Partial Response (PR) was defined as at least a 30% decrease in sum of longest diameter of target lesions compared to baseline or the complete disappearance of target lesions, with persistence of 1 or more nontarget lesion(s) and no new lesions.
Overall Survival | Time from randomization to death by any cause, assessed for up to 3 years
  Overall survival (OS) is the duration from date of randomization to date of death from any cause. Participants were censored at the date they were last known to be alive.

OTHER OUTCOMES:
Percentage of Participants Experiencing an Adverse Event (AE) | Up to 2 years
  An AE is defined as any untoward medical occurrence in a participant administered study treatment which does not necessarily have to have a causal relationship with this treatment. An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study treatment or protocol-specified procedure, whether or not considered related to the study treatment or protocol-specified procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jiexia Zhang, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided